CLINICAL TRIAL: NCT07125885
Title: Serological, Metabolomic, and Genomic Studies of Endocrine Disorders in Pregnancy
Brief Title: Gongji Pregnancy Endorine Cohort Study
Acronym: GREAT
Status: Recruiting | Type: Observational
Sponsor: Shanghai General Hospital, China (Other)
Responsible Party: Principal Investigator, Yufan Wang, Chief Physician, Professor, Shanghai General Hospital, China
Other Study IDs: 2022SQ506
Record Dates: First submitted 2025-07-12; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Gestatiaonl Diabetes Mellitus; Thyroid Disease Pregnancy; Hyperglycemia in Pregnant Diabetic Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Stool, Serum/Plasma, Urine, Placenta

SUMMARY:
To explore the relationship between genetic factors, lifestyle, and drug interventions and the occurrence, development, adverse pregnancy outcomes, and postpartum maternal-infant outcomes of gestational endocrine diseases.

DETAILED DESCRIPTION:
Time Perspective: Prospective and retrospective

ELIGIBILITY:
Inclusion Criteria:

* Women preparing for pregnancy or pregnant women or within 1 year after giving birth
* Age ≥ 18 years old
* Signed the informed consent form to voluntarily enroll in the management follow-up

Exclusion Criteria:

* Individuals who are unable to communicate normally and those who are unwilling to cooperate
* Pregnant women with severe organic diseases or mental illnesses
* Any condition deemed by the investigator to affect eligibility for the study

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: The study will include patients who receive routine prenatal care, delivery, and postpartum endocrinology follow-up at Shanghai General Hospital
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2043-12-31 (Estimated); Study Completion 2043-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite adverse maternal and neonatal outcomes associated with gestational endocrine disorders | From delivery (Day 0) through the initial birth hospitalization, assessed up to 14 days postpartum.
  Unit of Measure: Percentage of pregnancies with ≥ 1 event (%) Description: The composite will be coded as Yes/No. An event is counted if any of the following occurs: preeclampsia, cesarean delivery, premature rupture of membranes, placental abruption, preterm birth, congenital malformations, macrosomia, large for gestational age, small for gestational age, neonatal hypoglycemia, neonatal hyperbilirubinemia, neonatal respiratory distress syndrome, neonatal intensive care unit admission, obstetric trauma or still birth. Data abstracted from electronic medical records.
Postpartum glucose metabolism outcomes in patients with endocrine disorders in pregnancy | From 6 weeks postpartum through long-term follow-up, with assessments at 6 weeks and every 12 months thereafter, for ≥3 years and up to 40 years postpartum.
  Percentage of patients with diabetes mellitus (%) Postpartum glucose metabolism will be assessed using an oral glucose tolerance test (OGTT) to determine the incidence of diabetes mellitus. Data will be collected from blood tests and medical records.
Postpartum thyroid disease outcomes in patients with endocrine disorders in pregnancy | From 6 weeks postpartum through long-term follow-up, with assessments at 6 weeks and every 12 months thereafter, for ≥3 years and up to 40 years postpartum.
  Unit of Measure: Changes in serum thyroid-stimulating hormone (TSH), free triiodothyronine (FT3), and free thyroxine (FT4) levels (mU/L, pg/mL) Postpartum thyroid disease outcomes will be evaluated by measuring serum thyroid-stimulating hormone (TSH), free triiodothyronine (FT3), and free thyroxine (FT4) levels. Changes in these biomarkers will be used to assess thyroid function recovery or progression of thyroid dysfunction (e.g., hypothyroidism or hyperthyroidism) postpartum. These levels will be compared to baseline values, which include both pre-pregnancy and pregnancy-associated measurements. Data will be obtained from blood tests and medical records.

SECONDARY OUTCOMES:
Incidence of abnormal glucose metabolism in offspring of women with gestational endocrine diseases | From 6 weeks postpartum through long-term follow-up, with assessments at 6 weeks and every 12 months thereafter, for ≥3 years and up to 40 years postpartum.
  Unit of Measure: Cumulative incidence of abnormal glucose metabolism (%) Abnormal glucose metabolism in offspring will be measured by conducting oral glucose tolerance tests (OGTT) and/or HbA1c tests. Data will be collected from clinical records and blood tests.
Incidence of thyroid disorders in offspring of women with gestational endocrine diseases | From 6 weeks postpartum through long-term follow-up, with assessments at 6 weeks and every 12 months thereafter, for ≥3 years and up to 40 years postpartum.
  Unit of Measure: Percentage of offspring with thyroid disorders (%) Thyroid disorders in offspring will be diagnosed by measuring serum thyroid-stimulating hormone (TSH), free thyroxine (FT4), and free triiodothyronine (FT3) levels. Data will be obtained from blood tests and medical records.
Growth Abnormalities in Offspring of Women with Gestational Endocrine Diseases | From 6 weeks postpartum through long-term follow-up, with assessments at 6 weeks and every 12 months thereafter, for ≥3 years and up to 40 years postpartum.
  Unit of Measure: Body Mass Index (BMI) (kg/m²) Growth abnormalities in offspring will be assessed through anthropometric measurements including weight (kg) and height (m). BMI will be calculated using the formula: BMI = weight (kg) / height² (m²). Data will be collected from routine pediatric examinations and medical records.
Developmental abnormalities in offspring of women with gestational endocrine diseases | From 6 weeks postpartum through long-term follow-up, with assessments at 6 weeks and every 12 months thereafter, for ≥3 years and up to 40 years postpartum.
  Unit of Measure: Percentage of offspring with developmental abnormalities (%) Developmental abnormalities will be assessed through motor skills evaluations (e.g., fine and gross motor skills) and cognitive development assessments. Data will be collected from routine pediatric evaluations and medical records.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, China, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Time Frame: Data will be uploaded to Zenodo and shared, starting 9 months and ending 36 months following article publication